CLINICAL TRIAL: NCT00000432
Title: A Controlled Trial of a Primary and Secondary Program for Lyme Disease
Brief Title: Lyme Disease Prevention Program
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Matthew H. Liang, MD, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Purpose: Prevention
Other Study IDs: P60 AR36308 NIAMS-017; P60AR036308 (NIH)
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Lyme Disease; Tick-Borne Diseases
Keywords: Lyme disease; Education evaluation; Communicable disease control; Outcomes research; Tick-transmitted diseases
MeSH Terms: conditions — Lyme Disease; Tick-Borne Diseases

INTERVENTIONS:
Behavioral: Education about disease prevention

SUMMARY:
This is a large study of an educational program on Lyme disease prevention for passengers on ferry boats going to Nantucket Island during the period from Memorial Day until Labor Day. Some boats provide passengers with the experimental program and the other boats provide a "control" program that the researchers can compare to the experimental program. The experimental program uses live performances by entertainers to teach people about Lyme disease prevention, and also uses additional printed materials. People on the control boats receive education on injury prevention and road safety while bicycling, rollerblading, and using mopeds. The main result we will look for is Lyme disease identified by a followup survey and confirmed by reviewing medical records. We will also ask some people to take part in a smaller study of behavior change. In this study, we will ask people to complete forms on self-efficacy (a person's belief in his or her ability to reach a certain goal), their plans to take preventive steps, and actual prevention behaviors. We also ask participants who report doctor visits or illness to provide confirmation of their use of health services.

DETAILED DESCRIPTION:
This is a large, randomized trial of a Lyme disease primary prevention program for passengers on ferry boats going to Nantucket Island for the period from Memorial Day until Labor Day. Boats are randomized to experimental or control interventions.

The experimental intervention is a performance-based educational program on Lyme disease prevention, and uses supplemental materials. An entertainment troupe delivers the intervention using comedy, theater, and vaudevillian techniques. The entertainers present three shows in different locations on the boat. Each show is about 10 minutes and covers the severity and likelihood of acquiring Lyme disease and the benefits of tick avoidance and search and removal behaviors. When people on experimental boats enroll in the study they receive the following free materials: a wallet-sized tick ID card, a laminated shower card with tick-removal instructions, a map showing tick habitats, a tick-feeling card, and an educational pamphlet. Control boats do not have performers. Participants on control boats receive education on road safety and injury prevention from rollerblade, bicycle, and skateboard accidents.

We will collect baseline data at enrollment, including name, address, demographics, resident/visitor status, length of stay on island, frequency of exposure to tick areas, history of tick-transmitted disease, and exposure to intervention. We will enroll a random subsample of participants in a study of behavior, and will ask them additional questions on self-efficacy, intention to perform prevention behaviors and attitude about or social support for practicing prevention behaviors while on the island.

We will follow people in the behavioral subsample at 1 week to find out their actual behaviors. We will follow all subjects at 2 months to find out self-reported disease status. We ask persons reporting a visit to an M.D. for illness to mail a form to their physician for confirmation of diagnosis and to provide information about health-care use. The main outcome is Lyme disease. Intermediate outcomes include change in self-efficacy, behavioral intention, and health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Ferry passengers traveling to Nantucket Island

Exclusion Criteria:

* Foreign (non-U.S.) residence

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20000
Dates: Start 1997-04; Primary Completion 2001-03 (Actual); Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew H. Liang, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Steamship Authority ferry boats to Nantucket Island, Hyannis, Massachusetts, United States

REFERENCES:
- [Background] Shadick NA, Daltroy LH, Phillips CB, Liang US, Liang MH. Determinants of tick-avoidance behaviors in an endemic area for Lyme disease. Am J Prev Med. 1997 Jul-Aug;13(4):265-70. PMID 9236962
- [Background] Phillips CB, Liang MH, Sangha O, Wright EA, Fossel AH, Lew RA, Fossel KK, Shadick NA. Lyme disease and preventive behaviors in residents of Nantucket Island, Massachusetts. Am J Prev Med. 2001 Apr;20(3):219-24. doi: 10.1016/s0749-3797(00)00315-9. PMID 11275450